CLINICAL TRIAL: NCT04259450
Title: A Phase 1/2a Open Label, Multicenter Study to Access the Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of AFM24 in Patients With Advanced Solid Tumors
Brief Title: Study to Assess AFM24 in Advanced Solid Cancers
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Enrollment into expansion cohorts in Phase 2 part was terminated due to sponsor decision
Sponsor: Affimed GmbH (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AFM24-101
Record Dates: First submitted 2020-02-03; First posted 2020-02-06 (Actual); Results first posted 2024-08-29 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-06

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (10):
- Phase 1- 14 mg Cohort 1 (Experimental): Subjects, with tumors known to express EGFR, who received 14 milligram (mg) AFM24 on Day 1, Day 8, Day 15, and Day 22 of a 28-day cycle.
  Interventions: Drug: 14 mg AFM24
- Phase 1- 40 mg Cohort 2 (Experimental): Subjects, with tumors known to express EGFR, who received 40 milligram (mg) AFM24 on Day 1, Day 8, Day 15, and Day 22 of a 28-day cycle.
  Interventions: Drug: 40 mg AFM24
- Phase 1- 80 mg Cohort 3 (Experimental): Subjects, with tumors known to express EGFR, who received 80 milligram (mg) AFM24 on Day 1, Day 8, Day 15, and Day 22 of a 28-day cycle.
  Interventions: Drug: 80 mg AFM24
- Phase 1- 160 mg Cohort 4 (Experimental): Subjects, with tumors known to express EGFR, who received 160 milligram (mg) AFM24 on Day 1, Day 8, Day 15, and Day 22 of a 28-day cycle.
  Interventions: Drug: 160 mg AFM24
- Phase 1- 320 mg Cohort 5 (Experimental): Subjects, with tumors known to express EGFR, who received 320 milligram (mg) AFM24 on Day 1, Day 8, Day 15, and Day 22 of a 28-day cycle.
  Interventions: Drug: 320 mg AFM24
- Phase 1- 480 mg Cohort 6 (Experimental): Subjects, with tumors known to express EGFR, who received 480 milligram (mg) AFM24 on Day 1, Day 8, Day 15, and Day 22 of a 28-day cycle.
  Interventions: Drug: 480 mg AFM24
- Phase 1- 720 mg Cohort 7 (Experimental): Subjects, with tumors known to express EGFR, who received 720 milligram (mg) AFM24 on Day 1, Day 8, Day 15, and Day 22 of a 28-day cycle. A dose could be given over two days (split day dosing).
  Interventions: Drug: 720 mg AFM24
- Phase 2- CRC 480 mg Cohort A (Experimental): Subjects with microsatellite stable (MSS) colorectal cancer (CRC) with rat sarcoma gene (RAS) wild-type tumor expressing EGFR who received 480 milligram (mg) AFM24 weekly on Day 1, Day 8, Day 15, and Day 22 of a 28-day cycle. A dose could be given over two days (split day dosing).
  Interventions: Drug: 480 mg AFM24
- Phase 2- ccRCC 480 mg Cohort B (Experimental): Subjects with clear cell renal cell carcinoma (ccRCC) expressing EGFR who received 480 milligram (mg) AFM24 weekly on Day 1, Day 8, Day 15, and Day 22 of a 28-day cycle. A dose could be given over two days (split day dosing).
  Interventions: Drug: 480 mg AFM24
- Phase 2- NSCLC 480 mg Cohort C (Experimental): Subjects with advanced or metastatic (non-small cell lung cancer) NSCLC with an epidermal growth factor receptor (EGFR) mutation who received 480 milligram (mg) AFM24 weekly on Day 1, Day 8, Day 15, and Day 22 of a 28-day cycle. A dose could be given over two days (split day dosing).
  Interventions: Drug: 480 mg AFM24

INTERVENTIONS:
Drug: 14 mg AFM24 — 14 milligram AFM24 weekly on Day 1, Day 8, Day 15, and Day 22 of a 28-day cycle.
  Arms: Phase 1- 14 mg Cohort 1
Drug: 40 mg AFM24 — 40 milligram AFM24 weekly on Day 1, Day 8, Day 15, and Day 22 of a 28-day cycle.
  Arms: Phase 1- 40 mg Cohort 2
Drug: 80 mg AFM24 — 80 milligram AFM24 weekly on Day 1, Day 8, Day 15, and Day 22 of a 28-day cycle.
  Arms: Phase 1- 80 mg Cohort 3
Drug: 160 mg AFM24 — 160 milligram AFM24 weekly on Day 1, Day 8, Day 15, and Day 22 of a 28-day cycle.
  Arms: Phase 1- 160 mg Cohort 4
Drug: 320 mg AFM24 — 320 milligram AFM24 weekly on Day 1, Day 8, Day 15, and Day 22 of a 28-day cycle.
  Arms: Phase 1- 320 mg Cohort 5
Drug: 480 mg AFM24 — 480 milligram AFM24 weekly on Day 1, Day 8, Day 15, and Day 22 of a 28-day cycle.
  Arms: Phase 1- 480 mg Cohort 6; Phase 2- CRC 480 mg Cohort A; Phase 2- NSCLC 480 mg Cohort C; Phase 2- ccRCC 480 mg Cohort B
Drug: 720 mg AFM24 — 720 milligram AFM24 weekly on Day 1, Day 8, Day 15, and Day 22 of a 28-day cycle.
  Arms: Phase 1- 720 mg Cohort 7

SUMMARY:
AFM24-101 is a first in human Phase 1/2a open-label, non-randomized, multi-center, multiple ascending dose escalation/expansion study evaluating AFM24 as monotherapy in patients with advanced solid malignancies whose disease has progressed after treatment with previous anticancer therapies.

AFM24 is a tetravalent bispecific (anti-human EGFR x anti-human CD16A) innate immune cell engaging recombinant antibody being developed to target EGFR-expressing solid tumors and has been designed to specifically utilize the cytotoxic potential of the innate immune system, in particular natural killer cells and macrophages for the specific and efficient elimination of EGFR expressing cancer cells.

DETAILED DESCRIPTION:
There will be two parts to this study: a dose escalation phase (1) and a dose expansion phase (2a).

The aim of the dose escalation phase is to determine the maximum tolerated dose (MTD) and establish the recommended Phase 2a dose (RP2D).

The dose escalation phase will be followed by the dose expansion phase once the MTD/RP2D of AFM24 monotherapy has been determined. The dose expansion phase of the study using the MTD/P2D is intended to collect preliminary evidence of efficacy and to further confirm the safety of AFM24 as a monotherapy. The expansion phase will have 3 arms based on tumor type.

* Renal cell carcinoma(clear cell), failing standard of care (SoC) that includes TKIs and PD1 targeted therapy
* Non-small cell lung cancer (EGFR-mut), failing SoC TKIs
* Colorectal cancer, failing SOC chemotherapy, VEGF(R) and EGFR targeted antibodies

ELIGIBILITY:
Inclusion Criteria:

* Adequate organ function
* Phase 1: Histologically or cytologically confirmed advanced or metastatic solid malignancies that are known to express EGFR
* Phase 1: Previously treated with ≥ 1 lines of anticancer therapy and have documented disease progression during or after their most recent line of anticancer therapy. In addition, either there is no further SOC therapy for the patient or the remaining SOC therapies are deemed not appropriate for the patient by the Investigator.
* Phase 1: Patients must have at least one tumor site that is accessible to biopsy
* Phase 2a: Measurable disease per RECIST 1.1
* Phase 2a: Histologically confirmed advanced or metastatic EGFR+ malignancies for each expansion cohorts:
* Colorectal Cancer (MSS), KRAS-wildtype: disease has progressed after ≥ 2 prior lines of therapy which must have included oxaliplatin, fluoropyrimidine, bevacizumab, and an anti-EGFR therapy
* ccRCC: disease has progressed after ≥ 2 prior lines of therapy which must have included a TKI and a checkpoint inhibitor
* metastatic NSCLC, EGFRmut: disease has progressed on/after after ≥ 1 prior lines of therapy for advanced disease including ≥ 1 prior TKI approved for EGFR mut NSCLC

Exclusion Criteria:

* Treatment with systemic anticancer therapy within 4 weeks of the first dose of study drug (6 weeks if therapy was mitomycin C and/or nitrosoureas), or within 5 half-lives of the agent if half-life is known and it is shorter, before first dose of study drug. Anticancer therapies include cytotoxic chemotherapy, targeted inhibitors, and immunotherapies, but do not include hormonal therapy or radiotherapy.
* Radiation therapy within 2 weeks before 1st dose of study drug or unresolved toxicity from previous radiotherapy.
* History of any other malignancy known to be active, with the exception of completely removed in situ cervical intra-epithelial neoplasia, non-melanoma skin cancer, DCIS, early stage prostate cancer that has been adequately treated, and other cancers from which the patient has been disease free for 3 years or longer.
* Currently participating in a study and receiving study therapy, or participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2020-04-07 (Actual); Primary Completion 2023-07-12 (Actual); Study Completion 2024-06-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Emig, MD, Study Director — Affimed GmbH
Locations (13):
- United States (2):
  - University of Southern California, Los Angeles, California
  - Dana Faber Cancer Institute, Boston, Massachusetts
- Germany (3):
  - Nordwest Hospital GmbH, Frankfurt am Main, Hesse
  - University Duisburg-Essen, University Hospital Essen, Essen
  - University Hospital Hamburg-Eppendorf, Hamburg
- South Korea (3):
  - Seoul National University Bundang Hospital, Seongnam-si
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea St. Vincent's Hospital, Suwon
- Spain (4):
  - Vall d'Hebron Institute of Oncology, Barcelona
  - University Hospital Foundation Jimenez Diaz, Madrid
  - University Hospital HM Sanchinarro, Madrid
  - Hospital Clinic Universitario Biomedical Research institute INCLIVA, Valencia
- Institute of Cancer Research - Royal Marsden, London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was a phase 1/2a open-label, multicenter study to assess the safety, tolerability, pharmacokinetics and preliminary efficacy of AFM24 in patients with advanced solid cancers
Pre-assignment Details: Phase 1 subjects enrolled if they had a tumor known to express Epidermal Growth Factor Receptor (EGFR), Phase 2 subjects were screened for positive EGFR from tumor site. Specialists assessed the subjects, and they were enrolled in the study if they met all inclusion criteria and none of the exclusion criteria.
Period: Overall Study
Arm/Group | Phase 1- 14 mg Cohort 1 | Phase 1- 40 mg Cohort 2 | Phase 1- 80 mg Cohort 3 | Phase 1- 160 mg Cohort 4 | Phase 1- 320 mg Cohort 5 | Phase 1- 480 mg Cohort 6 | Phase 1- 720 mg Cohort 7 | Phase 2- CRC 480 mg Cohort A | Phase 2- ccRCC 480 mg Cohort B | Phase 2- NSCLC 480 mg Cohort C
Started | 2 | 6 | 4 | 5 | 6 | 6 | 6 | 19 | 8 | 23
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 2 | 6 | 4 | 5 | 6 | 6 | 6 | 19 | 8 | 23
Not completed — Adverse event/ Toxicity | 0 | 3 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 3
Not completed — Disease progression | 2 | 3 | 4 | 4 | 6 | 6 | 6 | 15 | 6 | 18
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Other than listed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2

BASELINE CHARACTERISTICS:
Population: Safety analysis set : consist of all subjects who received at least one dose of AFM24.
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 1- 14 mg Cohort 1 | Phase 1- 40 mg Cohort 2 | Phase 1- 80 mg Cohort 3 | Phase 1- 160 mg Cohort 4 | Phase 1- 320 mg Cohort 5 | Phase 1- 480 mg Cohort 6 | Phase 1- 720 mg Cohort 7 | Phase 2- CRC 480 mg Cohort A | Phase 2- ccRCC 480 mg Cohort B | Phase 2- NSCLC 480 mg Cohort C | Total
Number analyzed (Participants) | 2 | 6 | 4 | 5 | 6 | 6 | 6 | 19 | 8 | 23 | 85
Age, Continuous [Mean (Standard Deviation); unit: Years] | 73.0 (0.00) | 54.7 (14.12) | 47.3 (20.89) | 58.4 (11.35) | 57.7 (16.99) | 59.7 (12.08) | 53.8 (10.57) | 62.7 (9.32) | 67.1 (15.00) | 61.1 (11.83) | 60.2 (12.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 0 | 4 | 3 | 2 | 1 | 5 | 2 | 10 | 29
  Male | 1 | 5 | 4 | 1 | 3 | 4 | 5 | 14 | 6 | 13 | 56
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 1 | 2 | 1 | 0 | 0 | 1 | 1 | 1 | 9
  Not Hispanic or Latino | 2 | 2 | 3 | 3 | 5 | 6 | 6 | 18 | 7 | 21 | 73
  Unknown or Not Reported | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 10 | 1 | 18 | 32
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2
  White | 1 | 4 | 4 | 4 | 4 | 5 | 5 | 9 | 7 | 5 | 48
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Phase 1: The Number of Subjects With Dose Limiting Toxicities (DLTs) During Cycle 1
Description: The number of patients with dose limiting toxicities (DLTs) in the first cycle, as assessed by the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) v5.0. DLT is defined as an adverse event (AE) or abnormal laboratory value assessed as unrelated to underlying disease, disease progression, inter-current illness, or concomitant medications, that occurs ≤28 days following the first dose of AFM24 (Cycle 1).
Time Frame: During Cycle 1 (up to 28 days)
Population: The Dose-Determining Set (DDS): All patients in the safety set (all patients who received at least one dose of AFM24), who had either (a) experienced DLT at any time during Cycle 1, or (b) met the minimum safety evaluation requirements without experiencing DLT within Cycle 1.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1- 14 mg Cohort 1 | Phase 1- 40 mg Cohort 2 | Phase 1- 80 mg Cohort 3 | Phase 1- 160 mg Cohort 4 | Phase 1- 320 mg Cohort 5 | Phase 1- 480 mg Cohort 6 | Phase 1- 720 mg Cohort 7
Number analyzed (Participants) | 2 | 4 | 4 | 4 | 5 | 6 | 6
Participants | 0 | 1 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Phase 2a: Overall Response Rate (Complete Response [CR] + Partial Response [PR])
Description: Overall response as defined by achieving confirmed CR and/or PR assessed by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. Partial or complete response needs to be confirmed with repeated assessment at least 4 weeks after the initial assessment.
Time Frame: Up to approximately 16 weeks.
Population: The safety set: All patients who received at least one dose of AFM24.
Measure: Count of Participants; unit: Participants
Groups:
- Phase 2- CRC 480 mg Cohort A: Subjects with microsatellite stable (MSS) colorectal cancer (CRC) with rat sarcoma gene (RAS) wild-type tumor expressing EGFR who received 480 milligram (mg) AFM24 weekly on Day 1, Day 8, Day 15, and Day 22 of a 28-day cycle.
- Phase 2- ccRCC 480 mg Cohort B: Subjects with clear cell renal cell carcinoma (ccRCC) expressing EGFR who received 480 milligram (mg) AFM24 weekly on Day 1, Day 8, Day 15, and Day 22 of a 28-day cycle.
- Phase 2- NSCLC 480 mg Cohort C: Subjects with advanced or metastatic (non-small cell lung cancer) NSCLC with an epidermal growth factor receptor (EGFR) mutation who received 480 milligram (mg) AFM24 weekly on Day 1, Day 8, Day 15, and Day 22 of a 28-day cycle.
Arm/Group | Phase 2- CRC 480 mg Cohort A | Phase 2- ccRCC 480 mg Cohort B | Phase 2- NSCLC 480 mg Cohort C
Number analyzed (Participants) | 19 | 8 | 23
Participants | 0 | 0 | 2

3. Secondary Outcome: Phase 1: The Number of Subjects With Treatment-emergent Adverse Events (TEAEs)
Description: Adverse Events (AEs) will be summarized with patient counts by Medical Dictionary for Regulatory Activities (MedDRA) System Organ Classes (SOCs) and Preferred Terms (PTs).
Time Frame: From the start of first infusion till the last infusion + 30 days, up to approximately 43 weeks.
Population: The safety set: All patients who received at least one dose of AFM24.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1- 14 mg Cohort 1 | Phase 1- 40 mg Cohort 2 | Phase 1- 80 mg Cohort 3 | Phase 1- 160 mg Cohort 4 | Phase 1- 320 mg Cohort 5 | Phase 1- 480 mg Cohort 6 | Phase 1- 720 mg Cohort 7
Number analyzed (Participants) | 2 | 6 | 4 | 5 | 6 | 6 | 6
Participants | 2 | 6 | 4 | 5 | 6 | 6 | 6

4. Secondary Outcome: Phase 1: The Number of Subjects With Serious Adverse Events (SAEs)
Description: Serious adverse Events (SAEs) will be summarized with patient counts by Medical Dictionary for Regulatory Activities (MedDRA) System Organ Classes (SOCs) and Preferred Terms (PTs).
Time Frame: From the start of first infusion till the last infusion + 30 days, up to approximately 43 weeks.
Population: The safety set: All patients who received at least one dose of AFM24.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1- 14 mg Cohort 1 | Phase 1- 40 mg Cohort 2 | Phase 1- 80 mg Cohort 3 | Phase 1- 160 mg Cohort 4 | Phase 1- 320 mg Cohort 5 | Phase 1- 480 mg Cohort 6 | Phase 1- 720 mg Cohort 7
Number analyzed (Participants) | 2 | 6 | 4 | 5 | 6 | 6 | 6
Participants | 2 | 3 | 2 | 2 | 4 | 3 | 2

5. Secondary Outcome: Phase 1: Area Under the Concentration-time Curve From Time 0 to Time Tau (7 Days) of AFM24 in Plasma
Description: Area under the concentration-time curve from time 0 to time tau (7 days) of AFM24 in plasma (AUC0-168)
Time Frame: Pre-dose (2 hours maximum) and 15, 30, 45 min after start of infusion (SOI) and end of infusion (EOI) and 1, 4, 18, 24, 48, 144 hours after EOI on Cycle 1 Day 22.
Population: The Pharmacokinetic set: all subjects who received at least one adequately documented dose of study drug and had at least one adequately documented post dose pharmacokinetic (PK) measurement. Subjects were excluded if they did not have at least two quantifiable concentration values, two of which must have occurred after Tmax, this was the case for one subject in Cohort 6.
Measure: Mean (Standard Deviation); unit: hours*nanogram /milliLiter
Arm/Group | Phase 1- 14 mg Cohort 1 | Phase 1- 40 mg Cohort 2 | Phase 1- 80 mg Cohort 3 | Phase 1- 160 mg Cohort 4 | Phase 1- 320 mg Cohort 5 | Phase 1- 480 mg Cohort 6 | Phase 1- 720 mg Cohort 7
Number analyzed (Participants) | 2 | 3 | 4 | 4 | 6 | 5 | 6
hours*nanogram /milliLiter | 53400 (61700) | 549000 (254000) | 1290000 (395000) | 4940000 (1370000) | 18100000 (6120000) | 28700000 (7620000) | 40200000 (12000000)

6. Secondary Outcome: Phase 1: Maximum Plasma Concentration (Cmax) of AFM24
Description: Maximum measured concentration (Cmax) of AFM24 in plasma
Time Frame: Pre-dose (2 hours maximum) and 15, 30, 45 min after start of infusion (SOI) and end of infusion (EOI) and 1, 4, 18, 24, 48, 144 hours after EOI on Cycle 1 Day 1 and on pre-dose (2 hours maximum) Cycle 1 Day 8.
Population: The Pharmacokinetic set: all subjects who received at least one adequately documented dose of study drug and had at least one adequately documented post dose PK measurement.
Measure: Mean (Standard Deviation); unit: nanogram /milliLiter
Arm/Group | Phase 1- 14 mg Cohort 1 | Phase 1- 40 mg Cohort 2 | Phase 1- 80 mg Cohort 3 | Phase 1- 160 mg Cohort 4 | Phase 1- 320 mg Cohort 5 | Phase 1- 480 mg Cohort 6 | Phase 1- 720 mg Cohort 7
Number analyzed (Participants) | 2 | 3 | 4 | 4 | 6 | 6 | 6
nanogram /milliLiter | 3290 (2860) | 13200 (3100) | 29200 (6620) | 60900 (17600) | 204000 (55600) | 298000 (71100) | 354000 (104000)

7. Secondary Outcome: Phase 1: Time of Maximum Observed Concentration (Tmax) of AFM24
Description: First time to maximum observed concentration of AFM24 sampled during a dosing interval.
Time Frame: as for outcome 5
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Phase 1- 14 mg Cohort 1 | Phase 1- 40 mg Cohort 2 | Phase 1- 80 mg Cohort 3 | Phase 1- 160 mg Cohort 4 | Phase 1- 320 mg Cohort 5 | Phase 1- 480 mg Cohort 6 | Phase 1- 720 mg Cohort 7
Number analyzed (Participants) | 2 | 3 | 4 | 4 | 6 | 6 | 6
hours | 1.84 (1.19) | 3.43 (1.97) | 5.63 (1.71) | 5.64 (1.30) | 7.18 (0.564) | 7.52 (1.38) | 5.21 (0.280)

8. Secondary Outcome: Phase 1: Minimum Plasma Concentration (Cmin) of AFM24
Description: Minimum measured concentration (Cmin) of AFM24 in plasma
Time Frame: Pre-dose (2 hours maximum) and 15, 30, 45 min after start of infusion (SOI) and end of infusion (EOI) and 1, 4, 18, 24, 48, 144 hours after EOI on Cycle 1 Day 1 and on pre-dose (2 hours maximum) Cycle 1 Day 22.
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Phase 1- 14 mg Cohort 1 | Phase 1- 40 mg Cohort 2 | Phase 1- 80 mg Cohort 3 | Phase 1- 160 mg Cohort 4 | Phase 1- 320 mg Cohort 5 | Phase 1- 480 mg Cohort 6 | Phase 1- 720 mg Cohort 7
Number analyzed (Participants) | 2 | 3 | 4 | 4 | 6 | 6 | 6
ng/mL | 32.7 (46.2) | 311 (281) | 810 (482) | 12000 (3540) | 73800 (40600) | 117000 (49600) | 233000 (113000)

9. Secondary Outcome: Phase 1: The Number of Subjects Who Developed Anti-drug Antibodies (ADAs) and Neutralizing ADAs During Treatment With AFM24
Description: The number of subjects who developed anti-drug antibodies (ADAs) at any time during the study.
Time Frame: Pre-dose cycle 1 Day 1 and end of treatment, up to approximately 39 weeks.
Population: The safety set: All patients who received at least one dose of AFM24.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1- 14 mg Cohort 1 | Phase 1- 40 mg Cohort 2 | Phase 1- 80 mg Cohort 3 | Phase 1- 160 mg Cohort 4 | Phase 1- 320 mg Cohort 5 | Phase 1- 480 mg Cohort 6 | Phase 1- 720 mg Cohort 7
Number analyzed (Participants) | 2 | 6 | 4 | 5 | 6 | 6 | 6
Participants | 1 | 4 | 2 | 3 | 1 | 0 | 1

10. Secondary Outcome: Phase 1: Overall Response Rate (Complete Response (CR) + Partial Response (PR))
Description: Overall response as defined by achieving confirmed CR and/or PR assessed by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. Partial or complete response needs to be confirmed with repeated assessment at least 4 weeks after the initial assessment by local reader.
Time Frame: From the start of first infusion till the last infusion + 30 days, up to approximately 43 weeks.
Population: The safety set: All patients who received at least one dose of AFM24.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1- 14 mg Cohort 1 | Phase 1- 40 mg Cohort 2 | Phase 1- 80 mg Cohort 3 | Phase 1- 160 mg Cohort 4 | Phase 1- 320 mg Cohort 5 | Phase 1- 480 mg Cohort 6 | Phase 1- 720 mg Cohort 7
Number analyzed (Participants) | 2 | 6 | 4 | 5 | 6 | 6 | 6
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0

11. Secondary Outcome: Phase 1: Duration of Response Rate (DOR)
Description: The DOR defined as time from first assessment of partial response (PR) or complete response (CR) to follow-on first assessment of progressive disease will be summarized by descriptive statistics including median DOR and where appropriate the respective 95% confidence intervals (CIs).
Time Frame: through study completion (estimated up to 24 weeks)
Population: No subjects had a response.
Arm/Group | Phase 1- 14 mg Cohort 1 | Phase 1- 40 mg Cohort 2 | Phase 1- 80 mg Cohort 3 | Phase 1- 160 mg Cohort 4 | Phase 1- 320 mg Cohort 5 | Phase 1- 480 mg Cohort 6 | Phase 1- 720 mg Cohort 7
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

12. Secondary Outcome: Phase 1: Disease Control Rate (Complete Response (CR) + Partial Response (PR) +Stable Disease (SD))
Description: Disease control as defined by achieving CR and/or PR and/or SD assessed by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.
Time Frame: From the start of first infusion till the last infusion + 30 days, up to approximately 43 weeks.
Population: The safety set: All patients who received at least one dose of AFM24.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1- 14 mg Cohort 1 | Phase 1- 40 mg Cohort 2 | Phase 1- 80 mg Cohort 3 | Phase 1- 160 mg Cohort 4 | Phase 1- 320 mg Cohort 5 | Phase 1- 480 mg Cohort 6 | Phase 1- 720 mg Cohort 7
Number analyzed (Participants) | 2 | 6 | 4 | 5 | 6 | 6 | 6
Participants | 0 | 1 | 0 | 0 | 0 | 2 | 1

13. Secondary Outcome: Phase 2a: The Number of Subjects With Treatment-emergent Adverse Events (TEAEs)
Description: as for outcome 3
Time Frame: From the start of first infusion till the last infusion + 30 days, up to approximately 105 weeks.
Population: The safety set: All patients who received at least one dose of AFM24.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2- CRC 480 mg Cohort A | Phase 2- ccRCC 480 mg Cohort B | Phase 2- NSCLC 480 mg Cohort C
Number analyzed (Participants) | 19 | 8 | 23
Participants | 19 | 8 | 23

14. Secondary Outcome: Phase 2a: The Number of Subjects With Serious Adverse Events (SAEs)
Description: as for outcome 4
Time Frame: From the start of first infusion till the last infusion + 30 days, up to approximately 105 weeks.
Population: The safety set: All patients who received at least one dose of AFM24.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2- CRC 480 mg Cohort A | Phase 2- ccRCC 480 mg Cohort B | Phase 2- NSCLC 480 mg Cohort C
Number analyzed (Participants) | 19 | 8 | 23
Participants | 8 | 6 | 8

15. Secondary Outcome: Phase 2a: Trough Concentration (Ctrough) of AFM24
Description: Trough concentration (Ctrough) of AFM24 in plasma.
Time Frame: Pre-dose (2 hours maximum) on Cycle 1 Day 22.
Population: The safety set: All patients who received at least one dose of AFM24.
Measure: Mean (Standard Deviation); unit: ng/mL (nanogram/milliliter)
Arm/Group | Phase 2- CRC 480 mg Cohort A | Phase 2- ccRCC 480 mg Cohort B | Phase 2- NSCLC 480 mg Cohort C
Number analyzed (Participants) | 19 | 8 | 23
ng/mL (nanogram/milliliter) | 69155.7 (32573.34) | 77642.7 (79113.19) | 84616.7 (36176.09)

16. Secondary Outcome: Phase 2a: Maximum Plasma Concentration (Cmax) of AFM24
Description: Maximum measured concentration (Cmax) of AFM24 in plasma.
Time Frame: Pre-dose (2 hours maximum) on Cycle 1 Day 22 and at end of infusion (EOI) on Cycle 1 Day 22.
Population: The safety set: All patients who received at least one dose of AFM24.
Measure: Mean (Standard Deviation); unit: ng/mL (nanogram/milliliter)
Arm/Group | Phase 2- CRC 480 mg Cohort A | Phase 2- ccRCC 480 mg Cohort B | Phase 2- NSCLC 480 mg Cohort C
Number analyzed (Participants) | 19 | 8 | 23
ng/mL (nanogram/milliliter) | 254285.7 (145002.08) | 170428.6 (71327.55) | 272111.1 (111029.35)

17. Secondary Outcome: Phase 2a: The Number of Subjects Who Developed Anti-drug Antibodies (ADAs) During Treatment With AFM24
Description: The number of subjects who developed anti-drug antibodies (ADAs) at any time during the study.
Time Frame: Pre-dose cycle 1 Day 1 and end of treatment, up to approximately 101 weeks.
Population: The safety set: All patients who received at least one dose of AFM24.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2- CRC 480 mg Cohort A | Phase 2- ccRCC 480 mg Cohort B | Phase 2- NSCLC 480 mg Cohort C
Number analyzed (Participants) | 19 | 8 | 23
Participants | 3 | 1 | 8

18. Secondary Outcome: Phase 2a: Overall Response Rate (Complete Response [CR] + Partial Response [PR]) Assessed by Central RECIST v1.1
Description: Overall response as defined by achieving confirmed CR and/or PR assessed by Central Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. Partial or complete response needs to be confirmed with repeated assessment at least 4 weeks after the initial assessment.
Time Frame: From the start of first infusion till the last infusion + 30 days, up to approximately 105 weeks.
Population: The safety set: All patients who received at least one dose of AFM24.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2- CRC 480 mg Cohort A | Phase 2- ccRCC 480 mg Cohort B | Phase 2- NSCLC 480 mg Cohort C
Number analyzed (Participants) | 19 | 8 | 23
Participants | 0 | 0 | 0

19. Secondary Outcome: Phase 2a: Duration of Response Rate (DOR) by RECIST v1.1 by Local Review
Description: The DOR defined as time from first assessment of partial response (PR) or complete response (CR) to follow-on first assessment of progressive disease will be summarized by descriptive statistics including median DOR and where appropriate the respective 95% confidence intervals (CIs). Assessments by local reader used only.
Time Frame: From the start of first infusion till the last infusion + 30 days, up to approximately 105 weeks.
Population: All patients who received at least one dose of AFM24 and who had a response by RECIST v1.1 by Local Review.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 2- NSCLC 480 mg Cohort C | Phase 2- ccRCC 480 mg Cohort B | Phase 2- CRC 480 mg Cohort A
Number analyzed (Participants) | 2 | 0 | 0
Months | NA [3.61 to NA] — Not enough events to calculate the data. |  |

20. Secondary Outcome: Phase 2a: Duration of Response Rate (DOR) by RECIST v1.1 by Central Review
Description: The DOR defined as time from first assessment of partial response (PR) or complete response (CR) to follow-on first assessment of progressive disease will be summarized by descriptive statistics including median DOR and where appropriate the respective 95% confidence intervals (CIs). Assessment by central reader used only.
Time Frame: From the start of first infusion till the last infusion + 30 days, up to approximately 105 weeks.
Population: All patients who received at least one dose of AFM24 and who had a response by RECIST v1.1 by Central Review.
Arm/Group | Phase 2- NSCLC 480 mg Cohort C | Phase 2- ccRCC 480 mg Cohort B | Phase 2- CRC 480 mg Cohort A
Number analyzed (Participants) | 0 | 0 | 0

21. Secondary Outcome: Phase 2a: Disease Control Rate (Complete Response (CR) + Partial Response (PR) +Stable Disease (SD))
Description: Disease control as defined by achieving CR and/or PR and/or SD assessed by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. Disease control was assessed by local RECIST v1.1 and by central RECIST v1.1.
Time Frame: From the start of first infusion till the last infusion + 30 days, up to approximately 105 weeks.
Population: The safety set: All patients who received at least one dose of AFM24.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2- CRC 480 mg Cohort A | Phase 2- ccRCC 480 mg Cohort B | Phase 2- NSCLC 480 mg Cohort C
Number analyzed (Participants) | 19 | 8 | 23
Participants
  Local RECIST v1.1 | 2 | 2 | 9
  Central RECIST v1.1 | 1 | 0 | 2

22. Secondary Outcome: Phase 2a: Progression-free-survival (PFS)
Description: Progression-Free Survival (PFS) was defined as (date of first progression - date of first study drug injection)/30.4375. PFS was measured by local and central assessments.
Time Frame: From the start of first infusion till the last infusion + 30 days, up to approximately 105 weeks.
Population: The safety set: All patients who received at least one dose of AFM24.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 2- CRC 480 mg Cohort A | Phase 2- ccRCC 480 mg Cohort B | Phase 2- NSCLC 480 mg Cohort C
Number analyzed (Participants) | 19 | 8 | 23
Months
  Local RECIST v1.1 | 1.61 [1.15 to 1.64] | 2.55 [0.43 to NA] — Not enough events to calculate the data. | 3.68 [1.61 to 5.36]
  Central RECIST v1.1 | 3.88 [1.61 to 5.88] | 8.15 [0.43 to NA] — Not enough events to calculate the data. | 3.52 [1.54 to 10.68]

23. Secondary Outcome: Phase 2a: Overall Survival
Description: Overall Survival (OS) was defined as (date of death - date of first dose)/30.4375. Patients alive at the end of study will be censored on the last date of observation.
Time Frame: From the start of first infusion till the last infusion + 30 days, up to approximately 105 weeks.
Population: The safety set: All patients who received at least one dose of AFM24.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 2- CRC 480 mg Cohort A | Phase 2- ccRCC 480 mg Cohort B | Phase 2- NSCLC 480 mg Cohort C
Number analyzed (Participants) | 19 | 8 | 23
Months | 6.64 [3.88 to 10.71] | 8.87 [0.43 to NA] — Not enough events to calculate the data. | NA [9.26 to NA] — Not enough events to calculate the data.

ADVERSE EVENTS:
Time Frame: From the start of first infusion till the last infusion + 30 days, up to approximately 105 weeks
Description: The safety set consisted of all subjects who received at least one dose of AFM24.
Arm/Group | Phase 1- 14 mg Cohort 1 | Phase 1- 40 mg Cohort 2 | Phase 1- 80 mg Cohort 3 | Phase 1- 160 mg Cohort 4 | Phase 1- 320 mg Cohort 5 | Phase 1- 480 mg Cohort 6 | Phase 1- 720 mg Cohort 7 | Phase 2- CRC 480 mg Cohort A | Phase 2- ccRCC 480 mg Cohort B | Phase 2- NSCLC 480 mg Cohort C
All-Cause Mortality (participants affected / at risk) | 1/2 | 6/6 | 4/4 | 3/5 | 4/6 | 4/6 | 6/6 | 14/19 | 6/8 | 7/23
Serious Adverse Events (participants affected / at risk) | 2/2 | 3/6 | 2/4 | 2/5 | 4/6 | 3/6 | 2/6 | 8/19 | 6/8 | 8/23
Other Adverse Events (participants affected / at risk) | 2/2 | 5/6 | 4/4 | 5/5 | 6/6 | 6/6 | 6/6 | 19/19 | 8/8 | 22/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1- 14 mg Cohort 1 (N=2) | Phase 1- 40 mg Cohort 2 (N=6) | Phase 1- 80 mg Cohort 3 (N=4) | Phase 1- 160 mg Cohort 4 (N=5) | Phase 1- 320 mg Cohort 5 (N=6) | Phase 1- 480 mg Cohort 6 (N=6) | Phase 1- 720 mg Cohort 7 (N=6) | Phase 2- CRC 480 mg Cohort A (N=19) | Phase 2- ccRCC 480 mg Cohort B (N=8) | Phase 2- NSCLC 480 mg Cohort C (N=23)
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Cholangitis infective (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Failure to thrive (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blindness (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bile duct stenosis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dilatation intrahepatic duct acquired (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
COVID-19 pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oesophageal candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vascular device infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Anorectal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bacterial abscess central nervous system (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Epilepsy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urinary tract obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1- 14 mg Cohort 1 (N=2) | Phase 1- 40 mg Cohort 2 (N=6) | Phase 1- 80 mg Cohort 3 (N=4) | Phase 1- 160 mg Cohort 4 (N=5) | Phase 1- 320 mg Cohort 5 (N=6) | Phase 1- 480 mg Cohort 6 (N=6) | Phase 1- 720 mg Cohort 7 (N=6) | Phase 2- CRC 480 mg Cohort A (N=19) | Phase 2- ccRCC 480 mg Cohort B (N=8) | Phase 2- NSCLC 480 mg Cohort C (N=23)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (4) | 5 (42) | 3 (4) | 4 (5) | 3 (3) | 6 (9) | 4 (4) | 15 (18) | 5 (7) | 19 (26)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Radiation pneumonitis (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sunburn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 3 (7) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 3 (5) | 2 (4) | 1 (1) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 3 (7) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 2 (5) | 3 (4) | 1 (1) | 0 (0)
Blood pressure decreased (Investigations) | 0 (0) | 1 (15) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 1 (3) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 1 (2) | 1 (2) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 5 (7)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alpha tumour necrosis factor increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
C-reactive protein increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
International normalised ratio increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Serum ferritin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urine output decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (3) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 2 (2) | 4 (7) | 1 (1) | 2 (2) | 4 (4)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (3) | 3 (3) | 4 (5) | 3 (3) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 3 (6) | 2 (2) | 1 (1) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Defaecation urgency (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fistula of small intestine (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 4 (5) | 0 (0) | 3 (6) | 2 (2) | 3 (4) | 3 (3)
Pyrexia (General disorders) | 0 (0) | 1 (5) | 2 (3) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 4 (4) | 0 (0) | 2 (2)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 4 (4) | 2 (5) | 3 (4)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Feeling of body temperature change (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infusion site extravasation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Temperature regulation disorder (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (7) | 2 (12) | 1 (3) | 3 (5) | 1 (3) | 1 (3)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 2 (3) | 0 (0) | 1 (2) | 1 (3) | 0 (0) | 1 (1) | 4 (9) | 1 (1) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 4 (5) | 3 (5) | 1 (1) | 0 (0) | 3 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (3) | 4 (6) | 2 (2) | 3 (3)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (2) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 1 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 1 (3) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 2 (3)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Axillary mass (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Coccydynia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (5) | 1 (1) | 2 (2) | 0 (0) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 5 (6)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (3) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (2) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (2) | 0 (0) | 1 (3) | 4 (4)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 1 (2) | 1 (1) | 1 (2) | 1 (1) | 2 (3) | 3 (3)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 2 (2) | 1 (1) | 2 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aphasia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bell's palsy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Klebsiella urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Rash pustular (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vascular device infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 1 (3) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (3) | 1 (1) | 1 (1)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Chloropsia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Conjunctival haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diplopia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Halo vision (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acrochordon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cytokine release syndrome (Immune system disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic pain (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Jaundice (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hydrocele (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Testicular pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
The central review of scans was terminated prematurely.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor has the right to review communications for 90 days prior to public release (whereby the sponsor may ask to consider modifications to ensure necessary protection of sponsor's IP). Any publication shall be not made before the first multi-centre publication if the study is a part of a multi-centred clinical trial. Also, if a publication concerns the analyses of data from a multi-centred clinical trial, the communication shall make reference to the relevant multi-centre publication

DOCUMENTS (2):
  • Study Protocol (2023-07-26): https://cdn.clinicaltrials.gov/large-docs/50/NCT04259450/Prot_000.pdf
  • Statistical Analysis Plan (2023-01-27): https://cdn.clinicaltrials.gov/large-docs/50/NCT04259450/SAP_001.pdf